CLINICAL TRIAL: NCT07034495
Title: Comparing of Laparotomy, Laparoscopy, and daVinci in Whipple, Hepatectomy, Pancreatectomy, and Gastrectomy
Brief Title: Laparotomy, Laparoscopy, da Vinci System
Status: Completed | Type: Observational
Sponsor: National Chung Hsing University (Other)
Collaborators: Chung Shan Medical University (Other)
Responsible Party: Principal Investigator, LIN, Ming-Hung, Professor, National Chung Hsing University
Other Study IDs: CS1-20103
Record Dates: First submitted 2025-06-01; First posted 2025-06-24 (Actual); Last update posted 2025-06-24 (Actual); Status verified 2025-06

CONDITIONS: Stomach Neoplasms; Pancreatic Neoplasms; Liver Neoplasms; Periampullary Neoplasms; Cholangiocarcinoma; Chronic Pancreatitis; Benign Liver Tumors; Pancreatic Cysts
Keywords: Whipple; hepatectomy; pancreatectomy; gastrectomy robotic surger; da Vinci Xi
MeSH Terms: conditions — Stomach Neoplasms; Pancreatic Neoplasms; Liver Neoplasms; Cholangiocarcinoma; Pancreatitis, Chronic; Pancreatic Cyst

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 4 Weeks
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- three surgical methods in Laparotomy, Laparoscope, and da Vinci: no intervention

SUMMARY:
1. This study looks at whether newer surgical tools-like the da Vinci robotic system-can help patients recover better after major abdominal surgeries. It compares three surgery methods: traditional open surgery, standard laparoscopic (minimally invasive) surgery, and robotic surgery.
2. The research focused on four common operations: Stomach surgery (gastrectomy), Pancreas surgery (pancreatectomy), Liver surgery (hepatectomy) and andWhipple procedure
3. Researchers looked at medical records from 486 patients over five years. They compared how long each surgery took, how much blood was lost, and how many days patients stayed in the hospital.
4. The study wanted to see if robotic and laparoscopic surgeries help patients by making the surgery faster, safer, and with a quicker recovery.
5. The benefits depended on the type of surgery. In many cases, robotic and laparoscopic surgery led to shorter hospital stays, less bleeding, or faster surgeries. These results suggest that using newer technology can help make surgeries safer and recovery easier for patients.

DETAILED DESCRIPTION:
1. The study was conducted with the assistance of Chung Shan Medical University's MIS (Minimally Invasive Surgery) Center, which included the general surgery team with extensive experience in open surgery, laparoscopic surgery, and Da Vinci surgery. The study collected a five-year dataset of patients from July 2015 to September 2019 at Chung Shan Medical University Hospital. A total of 486 patients (mean age = 57.96 ± 15.71 years) were enrolled in this study, comprising 269 males (mean age = 58.39 ± 15.49 years) and 217 female patients (mean age = 57.48 ± 16.00 years). All patients underwent robotic surgery for gastrectomy, liver resection, or pancreatectomy during the study period.
2. Regardless of the surgical methods (laparotomy, laparoscopy, or da Vinci system), the first step after the patient enters the operating room is always anesthesia. After administering anesthesia, the following different operation procedures result in different viewing images. During laparotomy, the surgeon opens the patient's body directly and operates with the naked eye. One disadvantage of laparotomy is that large wounds require more time to recover. In 2-dimensional (2D) image laparoscopy, a 2D screen shows an image that allows the surgeon to perform stereoscopic surgery. Although most surgical processes are similar between laparoscopy and robotic surgery, the imaging system has undergone significant improvements in robotic surgery. In surgery using the da Vinci system, an endoscope that captures high-definition 3-dimensional (3D) images from the surgical site is utilized. Images are processed using a video processor in the vision cart and displayed on a 3D viewer and touchscreen.
3. Statistical analysis was performed using SPSS version 20.0. One-way ANOVA was used to analyze two or more variables, and statistical significance was set at p < 0.05. In this study, we analyzed the relationship between three different groups of surgical methods and three perioperative outcomes (operative time, hospital stay, and bleeding) in the context of four Hepato-Pancreato-Biliary Surgery (HPB) surgeries.

ELIGIBILITY:
Inclusion Criteria:

1. Adult patients (age ≥ 18 years)
2. Underwent one of the following surgeries: gastrectomy, liver resection, or pancreatectomy
3. Received surgery at Chung Shan Medical University Hospital between July 2015 and September 2019
4. Surgery performed by the general surgery team with experience in open, laparoscopic, and robotic (da Vinci) surgery
5. Surgical method included one of the following: open surgery (laparotomy), laparoscopic surgery, or robotic (da Vinci) surgery

Exclusion Criteria:

1. Patients who underwent surgeries outside the specified types (i.e., not gastrectomy, liver resection, or pancreatectomy)
2. Patients with incomplete or missing perioperative data (e.g., operative time, blood loss, or hospital stay)
3. Patients who underwent combined or staged surgical procedures unrelated to the HPB domain

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: A population that needs robotic surgery for gastrectomy, liver resection, or pancreatectomy
Sampling Method: Non-Probability Sample
Enrollment: 486 (Actual)
Dates: Start 2015-07-01 (Actual); Primary Completion 2019-09-30 (Actual); Study Completion 2019-09-30 (Actual)

PRIMARY OUTCOMES:
operative time | From entry into the operating room for anesthesia induction to completion of skin closure at the end of surgery (Day 1, intraoperative period), assessed over an estimated duration of up to 10 hours
  The duration of the operation
bleeding | From initiation of surgery (skin incision) to completion of wound closure during surgery (Day 1, intraoperative period), assessed over an estimated duration of up to 10 hours.
  The amount of intraoperative bleeding

SECONDARY OUTCOMES:
hospital stay | From the date of surgery to the date of hospital discharge, assessed up to 55 days postoperatively
  The postoperative recovery time

CONTACTS AND LOCATIONS:
Overall Officials: Cheng-Ming Peng, MD, Ph.D., Study Director — Department of Surgery, da Vinci Minimally Invasive Surgery Center, Chung Shan Medical University Hospital
Locations (1):
- Chung Shan Medical University Hospital, Taichung, Taiwan

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will not be shared due to privacy concerns and institutional policies that restrict the disclosure of patient-level data, even in de-identified form. Additionally, there is currently no plan or infrastructure in place for secure data sharing in accordance with applicable ethical and legal standards.